CLINICAL TRIAL: NCT03411265
Title: Retaining Opioid Users Entering Medication Assisted Treatment and Encouraging HCV/HIV Testing Through Active Patients Sharing Experiences and the Provision of Information About Infections -an electroNic-health Application
Brief Title: RETAIN: Retaining Opioid Users Entering Medication Assisted Treatment and Encouraging HCV/HIV Testing
Acronym: RETAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Theresa Winhusen, PhD, Principal Investigator, University of Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2017-1074-1
Record Dates: First submitted 2018-01-10; First posted 2018-01-26 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Opioid-Related Disorders; Opioid-use Disorder; Drug Addiction; Substance Use Disorders
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RETAIN (Experimental): Participants who meet criteria will receive the RETAIN self-administered, e-health application intervention.
  Interventions: Other: self-administered, e-health application

INTERVENTIONS:
Other: self-administered, e-health application — RETAIN is a self-administered, e-health application and includes short videos in which patients who are successfully engaged in MAT discuss what they wish they had known about MAT and its benefits when they started treatment. The intervention is designed to maximize "scalability" - the administration would entail handing an electronic device (e.g., tablet, laptop, etc.) to an individual who would then self-administer the intervention.

SUMMARY:
The purpose of this research study is to:

1. assess how well individuals entering medication assisted treatment like the RETAIN e-health application as measured by their feedback on the intervention.
2. test the impact of RETAIN on knowledge about medication-assisted treatment(MAT).
3. assess treatment retention rates in patients completing the RETAIN intervention.
4. test the impact of RETAIN on knowledge about HCV/HIV
5. test the impact of RETAIN on interest in being tested for HCV/HIV

DETAILED DESCRIPTION:
The pre-post study of RETAIN will: 1) assess the acceptability of RETAIN as measured by participant feedback about the intervention; 2) test the impact of RETAIN on knowledge about MAT, as measured by the MAT Knowledge Assessment; 3) assess MAT retention rates in patients completing the RETAIN intervention; 4) test the impact of RETAIN on knowledge about HCV/ HIV; 5) test the impact of RETAIN on interest in being tested for HCV/HIV.

The acceptability of RETAIN will be assessed with a feedback form which includes questions about how helpful the intervention was (scale of 1-4), what the patient liked most and least about the intervention, and any suggestions for improving it. The average (and standard deviation) for the rated helpfulness of the intervention will be derived and the qualitative data about what they liked most and least about the intervention and suggestions for improvement will be tabulated. Pre-/post-changes in the percent of correct knowledge assessment items (i.e., about MAT and HCV/HIV) and interest in HCV/HIV testing will be analyzed using a Wilcoxon signed-rank test. The 3- and 6-month retention rates for RETAIN participants will be compared, using Fisher's exact tests, to the overall treatment retention rates at 3- and 6- months for the UC Health MAT clinics as determined by the retrospective chart review.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. Starting MAT with methadone or suboxone or in MAT for less than 2 weeks;

   Exclusion Criteria:
3. Does not sign the "short form" consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2018-09-06 (Actual); Study Completion 2018-09-06 (Actual)

PRIMARY OUTCOMES:
treatment retention status after 3 months | 3 months
  To compare with retention rates for the overall MAT clinics and use in sample size calculations for potential follow-on trial

SECONDARY OUTCOMES:
treatment retention status after 6 months | 6 months
  To compare with retention rates for the overall MAT clinics and use in sample size
MAT Knowledge Assessment | Pre and Post Tests in E-Health App Day 1
  To test the impact of RETAIN on knowledge about MAT
The Injection-Related Infection and Treatment Survey (I-RITS) | Pre and Post Tests in E-Health App Day 1
  To test the impact of RETAIN on knowledge about HCV and HIV
Feedback on the RETAIN e-health application | Day 1
  feedback includes questions about how helpful the intervention was (scale of 1-4), what the patient liked most and least about the intervention, and any suggestions for improving it.

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Winhusen, PhD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati Addiction Sciences Division, Cincinnati, Ohio, United States